CLINICAL TRIAL: NCT06130293
Title: The Effect of Daily Executive Function Training in School-aged Children With Autism Spectrum Disorder
Brief Title: VR Executive Training of School-aged Children With ASD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Meng-Ting Chen, Assistant professor, National Taiwan Normal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202310HM006
Record Dates: First submitted 2023-11-06; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Executive Function of School-aged Children With ASD

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR training (Experimental): Using VR training. 40 minutes per session, one session per week, and a total 8 weeks.
  Interventions: Device: VR game intervention
- Waiting list group (No Intervention)

INTERVENTIONS:
Device: VR game intervention — Using self-paced VR game to train.
  Arms: VR training

SUMMARY:
Many studies support that children with autism spectrum disorder (ASD) show executive dysfunction. The applicant's NSC project report also indicated that in all areas in the behavior rating inventory of executive function, the second edition (BRIEF-2), including inhibit, self-monitor, shift, emotional control, initiate, working memory, plan/organize, task-monitor, and organization of materials, children in the typically developmental group showed better performance than children in the ASD group. The results also indicated that compared to the diagnosis of ASD, an executive function could be a better predictor of daily life adaptation. Similarly, more and more researchers put their efforts into executive training. However, the results are mixed. A meta-analysis showed that technology-based training can effectively improve the executive function of children with ASD. Children with ASD love game-like training as it provides friendly environments to children with ASD and induces less anxiety. The applicant, therefore, plans to develop a virtual reality executive function training program in the first year based on the applicant's previous experience with executive function training. The game will include the components of visual searching, reaction time, shift, planning, and working memory. At the end of the game, the game will provide visual feedback to the children to train in self-monitoring. In the second year, the applicant will conduct a randomized controlled trial to investigate the effectiveness of the training program. I plan to include 70 children with ASD and randomly assign them to either the executive training or control groups. Executive function and daily life adaptation will be the indexes of the effectiveness of the study.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with ASD by a qualified healthcare professional
* meeting the ASD criteria by using ADOS-2
* IQ higher than 80.

Exclusion Criteria:

* not meeting the ASD criteria by using ADOS-2.
* IQ lower than 80.
* comorbid physical and/or motor disabilities.
* comorbid mental disabilities except ADHD.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Questionnaire of executive function | Week 0 (pre-intervention), Week 9 (post-intervention), and follow-up (Week 18 to Week 26)
  parent's and teacher's forms

SECONDARY OUTCOMES:
Questionnaire of adaptive behaviors | Week 0 (pre-intervention), Week 9 (post-intervention), and follow-up (Week 18 to Week 26)
  parent's and teacher's forms

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Normal University, Taipei, State, Taiwan

IPD SHARING:
Plan to Share IPD: No